CLINICAL TRIAL: NCT00628433
Title: A Phase I/II, Double-Blind, Randomized, Placebo-Controlled, Dose Ranging Study of the Safety, Tolerance, Pharmacokinetics and Activity of HE3286 When Administered Orally to Patients With Active, Mild-to-Moderate Ulcerative Colitis
Brief Title: Safety and Pharmacokinetics Study of HE3286 in Patients With Active, Mild-to-Moderate Ulcerative Colitis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Harbor Therapeutics (Industry)
Responsible Party: Nanette Onizuka-Handa, Sr. Vice President, Regulatory Affairs and Quality, Hollis-Eden Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HE3286-0301
Record Dates: First submitted 2008-02-25; First posted 2008-03-05 (Estimated); Last update posted 2011-06-14 (Estimated); Status verified 2011-06

CONDITIONS: Ulcerative Colitis
Keywords: phase I/II; ulcerative colitis; safety; tolerance; pharmacokinetics
MeSH Terms: conditions — Colitis, Ulcerative | interventions — 17-ethynyl-5-androstene-3, 7, 17-triol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- 2 (Experimental): HE3286 5 mg daily
  Interventions: Drug: HE3286
- 3 (Experimental): HE3286 10 mg daily
  Interventions: Drug: HE3286
- 4 (Experimental): HE3286 20 mg daily
  Interventions: Drug: HE3286
- 5 (Experimental): HE3286 4 mg daily
  Interventions: Drug: HE3286

INTERVENTIONS:
Drug: Placebo — Placebo
  Arms: 1
Drug: HE3286 — daily for 28 days
  Other Names: Triolex
  Arms: 2; 3; 4; 5

SUMMARY:
The purpose of this pilot, exploratory study is to evaluate the safety, tolerance, pharmacokinetics and potential activity of an investigational agent, HE3286, when administered orally, daily for 28 days to patients with mild-to-moderate ulcerative colitis.

DETAILED DESCRIPTION:
HE3286 has a potentially new mechanism of action that may improve the current therapeutic options available to patients with ulcerative colitis. In preclinical experiments, HE3286 has shown activity in animal models of ulcerative colitis. Additionally, HE3286 has shown to have anti-inflammatory activity associated with corticosteroids but without the side effects associated with corticosteroid use, such as immune suppression and bone loss.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age
* Diagnosed (> 6 weeks) or recently relapsed active mild-to-moderate ulcerative colitis based on colonoscopy or flexible sigmoidoscopy
* Mayo Scoring System for Assessment of Ulcerative Colitis Activity score of 4-9
* Stable dose prior to screening of 6-mercaptopurine (50-150 mg/day 6-MP) [at least 2 months], Azathioprine (50-100 mg/day) [at least 2 months], and 5-ASA [at least 2 weeks]
* For females of reproductive potential, agree to avoid pregnancy during the study and for 3 months following study completion, have a negative serum pregnancy test (b-HCG) at screening and negative urine pregnancy test and use an acceptable method of birth control
* No history of narcotic and/or alcohol abuse within 2 years of screening and agrees to consume < 6 oz. of wine or equivalent per day
* No experienced renal or liver disease by history and/or based on laboratory results
* Must provide voluntary, written, informed consent prior to screening evaluations and be able to follow verbal and written instructions
* Must be able to swallow capsules

Exclusion Criteria:

* Primary sclerosing cholangitis
* Positive for C. difficile toxin in the stool
* Requires hospitalization for treatment of severe ulcerative colitis
* History of clinically significant cardiovascular disease (including coronary artery disease), clinically significant hepatic, respiratory or renal abnormalities, or clinically significant endocrine disorders (not including diabetes)
* Clinically significant abnormalities on laboratory results (renal insufficiency, liver function abnormalities, abnormal WBC or ANC)
* Any clinically significant unstable medical abnormality, chronic disease, or active, serious clinical infection or condition, other than ulcerative colitis
* Uncontrolled hypertension defined as systolic BP > 160 mmHg and/or diastolic BP > 100 mmHg on three or more assessment on more than one day(blood pressure must be stable for > 3 months prior to screening)
* Malignancy within the past 5 years, except for successfully treated basal cell carcinoma of the skin
* Requiring or receiving anti-TNF-a or other immune modulating drugs (other than 6-MP or azathioprine) within 8 weeks prior to screening
* Requiring or receiving any of the following within 4 weeks of the screening visit: interleukins, steroids (i.e., anabolic steroids, glucocorticoids), narcotics, anti-cancer chemotherapeutic agents, metabolic inhibitors or nutraceuticals with immune enhancement claims
* Requiring oral or intravenous cortisone
* Requiring corticosteroid enemas
* Acute illness within 10 days prior to Day 1 or taking antibiotics for UC (but not for a infectious disease) within 14 days of Day 1
* Any clinical condition or receiving therapy that, in the opinion of the Investigator, would make the patient unsuitable for study or unable to comply with the dosing requirements

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2008-02; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
safety and pharmacokinetics | duration of the study

SECONDARY OUTCOMES:
assess activity on the signs and symptoms of active mild-to-moderate ulcerative colitis | duration of the study

CONTACTS AND LOCATIONS:
Overall Officials: Dwight R Stickney, MD, Principal Investigator — Harbor Therapeutics
Locations (9):
- United States (9):
  - Tucson, Arizona
  - Anaheim, California
  - Fresno, California
  - La Jolla, California
  - Denver, Colorado
  - Winter Park, Florida
  - Atlanta, Georgia
  - Louisville, Kentucky
  - El Paso, Texas